CLINICAL TRIAL: NCT05623826
Title: Feasibility and Efficacy of Imager, a Digital Training Intervention to Increase Reward Sensitivity: A Randomised Controlled Trial
Brief Title: Feasibility and Efficacy of a Digital Training Intervention to Increase Reward Sensitivity- Imager
Acronym: IMAGER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Johannes Gutenberg University Mainz (Other); Radboud University Medical Center (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UZH_Imager
Record Dates: First submitted 2022-04-25; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Stress
Keywords: stress; health; resilience

STUDY DESIGN:
Intervention Model Description: Parallel group design with control group completing only EMA, not EMI
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are informed of the two group design, individual group allocation is released to participants at the end of the study participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental (receiving EMA and Imager EMI)
  Interventions: Other: Cognitive- behavioral imagery-based training
- Control (No Intervention): Control (receiving EMA only)

INTERVENTIONS:
Other: Cognitive- behavioral imagery-based training — The EMI developed and tested here is based on theoretical and empirical findings and consists of several items and a repeated training using various individual scenarios from participants' life that will be presented to participants via an app on their smartphones.
  Other Names: Imager
  Arms: Experimental

SUMMARY:
Development and feasibility test of an Ecological Momentary Intervention (EMI) - Imager, to promote and improve stress resilience, specifically to increase reward sensitivity.

DETAILED DESCRIPTION:
Aim of the current project is to develop and test Ecological Momentary Intervention (EMI) - Imager, to promote and improve stress resilience, specifically to increase reward sensitivity. EMIs are mostly smartphone-based applications that deliver interventions to people as they go about in their daily lives. The EMI developed and tested here is based on theoretical and empirical findings and consists of several items and a repeated training using various individual scenarios from participants' life that will be presented to participants via an app on their smartphones.

This study tests the feasibility and effects of the EMI on a change in (i) reward sensitivity, (ii) mental imagery, and (iii) indices of perceived stress. One hundred twenty healthy student participants, aged 18-29 will be included in the study. Participants will be screened first and included if they score 5 points or more on the Reward Sensitivity Subscale of Behavioral Avoidance/Inhibition (BIS/BAS) scales. This is necessary in order to avoid a ceiling effect. Then, participants will be randomly assigned to an experimental (reward sensitivity EMI) or two of the control conditions (control EMA or waitlist). The reward sensitivity EMI group will be taught about experiencing rewards in daily life and will be asked to apply the specific techniques to personal situations repeatedly. The control EMA group will use the same app consisting of Ecological Momentary Assessment only, and the waitlist group will not receive any mobile app.

The training will last seven consecutive days and the app will send (i) 10 prompts per day to ask about the current mood of the user in control EMA and experimental groups and (ii) three prompts per day resulting in a total of 21 reward training sessions only in the experimental group. Participants will be able to use a special button triggering the intervention or EMA by themselves too. After one week, participants will return to the lab, fill in questionnaires and participate in behavioral tasks.

ELIGIBILITY:
Inclusion Criteria:

* being a student
* having sufficient knowledge of the German language
* being a smartphone user
* score of 5 points or more in Reward Sensitivity Subscale of Behavioral Avoidance/Inhibition (BIS/BAS) scales

Exclusion Criteria:

* having a mental illness or attending the psychotherapy

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2020-09-27 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Behavioural avoidance/inhibition (BIS/BAS) scales | one week: Pre- to post-intervention/control
  Self-reported reward sensitivity, scale range [0-15], higher score = worse outcome
The Sensitivity to Punishment and Sensitivity to Reward Questionnaire (SPSRQ) | one week: Pre- to post-intervention/control
  Self-reported reward sensitivity, scale range [0-24], higher score = better outcome
Perceived Stress Scale (PSS) | one week: Pre- to post-intervention/control
  Self-reported level of stress, scale range [0-40], higher score = worse outcome
Beck Depression Inventory II (BDI-II) | one week: Pre- to post-intervention/control
  Self-reported depressive symptoms, scale range [0-63], higher score = worse outcome
State-Trait Anxiety Inventory (STAI) | one week: Pre- to post-intervention/control
  Self-reported anxiety symptoms, scale range [20-80], higher score = worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Kleim, PhD, Principal Investigator — University of Zurich
Locations (1):
- Psychiatric University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Github, OSF
Supporting Information: CSR
Time Frame: from June 2022 onwards
Access Criteria: open to everyone